CLINICAL TRIAL: NCT05688501
Title: Development of a New Reliable, Easy and Reproducible Clinical-biological Scale Allowing to Select Patients Consulting in the Emergency Department for Upper Gastrointestinal Bleeding
Brief Title: Clinical-biological Score for Upper Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, Professor, Hôpital Universitaire Sahloul
Other Study IDs: GIB-ED
Record Dates: First submitted 2022-11-29; First posted 2023-01-18 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Gastro Intestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptiv group — no intervention

SUMMARY:
Gastrointestinal bleeding is a frequent reason for consultation in the Emergency Department. It is a real emergency associated with fairly significant morbidity and mortality.

The incidence of upper gastrointestinal bleeding (HDH) has been reported to be 67-103 per 100,000 adults per year in the UK with mortality rates of 2%-8%.

While Lower Gastrointestinal Bleeding (LBHB) has a lower incidence estimated at 33 per 100,000 adults per year. Additionally, compared to HDB, HDB appears to have less need for hemostatic intervention and lower mortality.

DETAILED DESCRIPTION:
Gastrointestinal bleeding is a frequent reason for consultation in the Emergency Department. It is a real emergency associated with fairly significant morbidity and mortality.

The incidence of upper gastrointestinal bleeding (HDH) has been reported to be 67-103 per 100,000 adults per year in the UK with mortality rates of 2%-8%.

While Lower Gastrointestinal Bleeding (LBHB) has a lower incidence estimated at 33 per 100,000 adults per year. Additionally, compared to HDB, HDB appears to have less need for hemostatic intervention and lower mortality.

Despite a decrease in incidence, the first cause of upper gastrointestinal bleeding remains peptic ulcer. That of lower digestive hemorrhage is diverticular hemorrhage, the incidence of which increases with the aging of the population.

Over time, the overall management of these haemorrhages has improved, in particular with better availability of endoscopic exploration from the emergency room consultation. However, the average time for digestive endoscopy was reported at 16 hours in a North African study published in 2012. Measures should be put in place to further improve access to endoscopy services for these patients, being given that a fifth of them received this care with delays exceeding 48 to 72 hours.

The indication of endoscopic exploration and its delay comes up against various practical difficulties. Hence the assessment of severity and the progressive risk of aggravation is essential for the emergency physician. Several prognostic or predictive clinical scores for worsening have been proposed. These scores remain underused and rarely applied to support and guide the therapeutic strategy.

These published prognostic scores aim to determine the risk of mortality, recurrence of bleeding and to identify patients requiring hospital treatment (transfusion, endoscopic or surgical treatment). Their interest lies in their ability to identify high-risk patients, for whom aggressive management is required, as well as low-risk patients for whom management could be delayed.

Indeed, in Tunisia, as for the vast majority of developing countries, one of the problems posed by the management of HDH remains the hospitalization of a majority of patients for monitoring, while only 1928% of between them will develop complications. These scores could be of great help in supporting and guiding the therapeutic strategy.

Among the predictive scores, it was found that "The Glasgow-Blatchford score", which is specific only to HDH and which aims to determine which patients are "low risk" and therefore candidates for outpatient management. Another score, the Rockall score, stratifies the risk of re-bleeding and death but requires endoscopic data provided by an emergency examination. These data remain missing in most cases, at least during the first hours of patient care.

Regardless of the source of bleeding, early identification of patients at high risk of mortality could allow targeted management, including specialist care and early interventions that may improve outcomes. At the other end of the spectrum, patients identified as being at very low risk of complications may benefit from less intensive management, which would help target resources to the appropriate patients.

Recent international recommendations concerning the management of these patients recommend the use of these scores in the emergency department for risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 consulting the emergency department of Sahloul Hospital in Sousse for exteriorized upper and/or lower digestive haemorrhage, of non-traumatic cause;

Exclusion Criteria:

* patient under the age of 18
* diagnosis of external hemorrhoids / perianal lesions
* Not consenting
* The lost sight

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Upper gastrointestinal bleeding (HDH) was defined as a presentation with hematemesis, blackish vomiting and/or melena.
  Lower gastrointestinal hemorrhage (LBH) was defined as a presentation with red blood or blood clots or blood mixed with stool on clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
re-bleeding | 30 days
  Hemorrhagic recurrence is defined by recurrence of hematemesis, melena or rectal bleeding after discharge from hospital within 30 days
re-hospitalization | 30 days
  re- hospitalisation for Hemorrhagic recurrence is defined by recurrence of hematemesis, melena or rectal bleeding after discharge from hospital within 30 days
All cause mortality | 30 days
  The primary outcome was all-cause in-hospital mortality rate
comparaison with the glasgow blatchford score | 30 days
  comparaison with the glasgow blatchford score

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Boukef, professor, Principal Investigator — CHU Sahloul, Emergency department, sousse
Locations (1):
- HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
after publication of the article